CLINICAL TRIAL: NCT04627597
Title: Informed Pre-operative Consent: Are We There Yet?
Brief Title: Patients' Comprehension and Internalization of Operative Consent Form
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/2638
Record Dates: First submitted 2020-10-23; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Informed Consent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective pilot study conducted within otolaryngology (ENT) clinics in a tertiary hospital between July and December 2016. 22 patients planned for common elective ENT operations were given a self-administered one-page survey on the same day after preoperative counselling. The investigators aim to identify if there are any associations between perceived and actual understanding of information given during pre-operative counselling and patient satisfaction with the process.

DETAILED DESCRIPTION:
As above and in later sections.

ELIGIBILITY:
Inclusion Criteria:

* Planned for common elective ENT operations
* English-speaking
* Unaccompanied
* Counselled with the use of a structured surgery-specific consent form

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients planned for common elective ENT operations in a tertiary hospital between July and December 2016
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Patient's perceived understanding of information given during pre-operative counselling (nominal score on questionnaire) | Through study completion, up to 6 months
  The score of how certain patients feel about information given during pre-operative counselling, as indicated on a self-administered questionnaire on the same day after pre-operative counselling
Patient's actual understanding of information given during pre-operative counselling (numeric score on questionnaire) | Through study completion, up to 6 months
  The score of correct answers patients give to factual questions about their surgery, as indicated on a self-administered questionnaire on the same day after pre-operative counselling
Patient's satisfaction with pre-operative counselling (nominal score on questionnaire) | Through study completion, up to 6 months
  The score of how satisfied patients are with pre-operative counselling, as indicated on a self-administered questionnaire on the same day after pre-operative counselling

CONTACTS AND LOCATIONS:
Overall Officials: Tze Choong Charn, MRCS, Principal Investigator — Singhealth Foundation

IPD SHARING:
Plan to Share IPD: No